CLINICAL TRIAL: NCT07018297
Title: Early Discharge With Subcutaneous Furosemide Versus Standard Care in Acute Heart Failure: A Cluster-Randomized Crossover Non-Inferiority Trial
Brief Title: Early Discharge With Subcutaneous Furosemide Versus Standard Care in Acute Heart Failure
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU2025-0766
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Acute Decompensated Heart Failure
Keywords: Subcutaneous Furosemide; Length of Stay (LOS); Hospitalization; Resource Allocation
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: Randomization at the cluster level (hospitalist subgroups, academic teaching teams, and cardiology practice groups). Each participating cluster will implement either the early discharge strategy or standard care for initial two-month blocks, followed by a crossover to the alternate strategy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early Discharge with Subcutaneous Furosemide (Experimental): The practice group randomized to early discharge with subcutaneous furosemide home infusion will begin initiation of subcutaneous furosemide (LASIX-ONYU) with a SQIN-Infusor device prior to discharge from the hospital. Dosing will be based on pre-admission oral furosemide requirements. Those with a home dose of ≤80mg/day oral furosemide will receive 80mg subcutaneous once daily at home and those with >80mg/day oral furosemide will receive 80mg subcutaneous twice daily at home.
  Interventions: Combination Product: Early Discharge with Lasix® ONYU (furosemide injection, for subcutaneous use) using SQIN-Infusor
- Usual Care (No Intervention): Usual inpatient care with IV furosemide. Discharge timing determined by treating physician per standard practice.

INTERVENTIONS:
Combination Product: Early Discharge with Lasix® ONYU (furosemide injection, for subcutaneous use) using SQIN-Infusor — Each practice group randomized to early discharge with subcutaneous furosemide will provide the patient with prefilled units of Lasix® ONYU furosemide injection containing 80 mg per 2.67 mL in a single-dose prefilled cartridge co-packaged with a single-use Disposable Unit of the Infusor that will be used in conjunction with the reusable unit of the Lasix ONYU Infusor. Dosing based on pre-admission oral furosemide requirements: ≤80mg/day oral furosemide will be given 80mg subcutaneous once daily or >80mg/day oral furosemide will be given 80mg subcutaneous twice daily. Dosing will be continued until clinical euvolemia is reached.
  Other Names: subcutaneous furosemide
  Arms: Early Discharge with Subcutaneous Furosemide

SUMMARY:
This will be a prospective, cluster-randomized, crossover, non-inferiority trial of 250 participants within 48 hours of an inpatient admission for heart failure or emergency department presentation for heart failure with plans for admission or observation/short-stay hospitalization comparing early discharge using subcutaneous furosemide to standard inpatient care. Individual practice groups will serve as "clusters" and the unit of randomization. Each participating cluster will implement either the early discharge strategy using the intervention or standard care for initial two-month blocks, followed by a crossover to the alternate strategy. The primary outcome is days alive and out of hospital at 30 days.

DETAILED DESCRIPTION:
HF contributes to over 1 million emergency department visits and nearly 1 million hospitalizations annually. The estimated annual mean cost per person with HF was $32,955 in 2017-2018, with the majority of costs due to hospitalization. The current standard of care typically involves admission for intravenous (IV) diuretics, monitoring for adequate decongestion, transition to oral diuretics, and discharge once clinical stability is achieved. The median length of stay for HF hospitalizations in the United States is 5 days but varies significantly across health systems and at the patient level. Extended hospitalizations, while traditionally considered necessary for complete decongestion, carry substantial risks, including increased risk of all-cause death and readmission. Patients experience deconditioning and increased frailty and are at risk for hospital-acquired complications, including infections, falls, and cognitive decline. Furthermore, prolonged hospitalization can lead to post-hospital syndrome, characterized by increased vulnerability and risk for adverse events in the immediate post-discharge period. For these reasons, reducing length of stay has emerged as a critical goal in HF management, aimed at both decreasing costs and improving patient outcomes by minimizing hospital-related complications and preserving quality of life.

Recent developments in subcutaneous furosemide formulations offer a potential solution to this clinical challenge. Pharmacokinetic studies demonstrate that subcutaneous furosemide achieves bioavailability comparable to IV administration and superior to oral formulations. The consistent absorption profile and reliable bioavailability of subcutaneous furosemide, combined with its ease of administration, presents an opportunity to provide hospital-level diuresis in the outpatient setting. This could enable earlier discharge while maintaining the intensity of diuretic therapy needed for complete decongestion. However, a critical knowledge gap exists regarding the safety and efficacy of an early discharge strategy utilizing subcutaneous furosemide compared to traditional inpatient management.

This trial aims to address this knowledge gap through a cluster-randomized crossover study comparing early discharge with subcutaneous furosemide to standard inpatient care and receipt of IV furosemide. By implementing standardized protocols across two major health systems, the investigators will evaluate whether this novel approach can safely reduce length of stay while maintaining clinical outcomes. The study design accounts for institutional variations in care delivery while providing robust data on safety, efficacy, and resource utilization. Results from this trial could fundamentally change the management paradigm for acute heart failure hospitalizations, potentially improving both healthcare efficiency and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Within 48 hours of inpatient stay OR ED presentation for HF with plans for admission OR observation stay/short-stay hospitalization for HF
* Expected to require at least 24 additional hours of IV diuretics
* Adequate home environment for self-care
* Patient or caregiver capable of operating subcutaneous delivery device

Exclusion Criteria:

* Cognitive impairment preventing informed consent
* Geographic barriers to follow-up
* Pregnancy or breastfeeding
* IV furosemide requirement >250mg/day
* eGFR <20 mL/min/1.73m2
* Type 1 myocardial infarction during index admission
* End-stage HF with receipt or consideration of heart transplant or LVAD or requiring inotropic or mechanical circulatory support
* Potassium <3.0 or >6.0 mmol/L or sodium <125 mmol/L

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of the hospital | 30-day
  Days alive and out of the hospital will be ascertained via retrospective review of the electronic health record.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 14-day, and 30-day. The Kansas City Cardiomyopathy Questionnaire Overall Summary Score ranges from 0-100, where 0 is worst quality of life and 100 is best quality of life.
  Longitudinal analysis of Kansas City Cardiomyopathy Overall Summary Scores
Change in N-terminal pro B-type natriuretic peptide | Baseline, 14-day, and 30-day
  Longitudinal analysis of N-terminal pro B-type natriuretic peptide (NT-proBNP) levels
Time-to-event for mortality and readmission | 30-day
  Time-to-event analyses for mortality and readmission outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott and White Health System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozkurt B, Ahmad T, Alexander KM, Baker WL, Bosak K, Breathett K, Fonarow GC, Heidenreich P, Ho JE, Hsich E, Ibrahim NE, Jones LM, Khan SS, Khazanie P, Koelling T, Krumholz HM, Khush KK, Lee C, Morris AA, Page RL 2nd, Pandey A, Piano MR, Stehlik J, Stevenson LW, Teerlink JR, Vaduganathan M, Ziaeian B; Writing Committee Members. Heart Failure Epidemiology and Outcomes Statistics: A Report of the Heart Failure Society of America. J Card Fail. 2023 Oct;29(10):1412-1451. doi: 10.1016/j.cardfail.2023.07.006. Epub 2023 Sep 26. No abstract available. PMID 37797885
- [Background] Bhatnagar R, Fonarow GC, Heidenreich PA, Ziaeian B. Expenditure on Heart Failure in the United States: The Medical Expenditure Panel Survey 2009-2018. JACC Heart Fail. 2022 Aug;10(8):571-580. doi: 10.1016/j.jchf.2022.05.006. Epub 2022 Jul 6. PMID 35902161
- [Background] Akintoye E, Briasoulis A, Egbe A, Adegbala O, Sheikh M, Singh M, Alliu S, Ahmed A, Asleh R, Kushwaha S, Levine D. Regional Variation in Mortality, Length of Stay, Cost, and Discharge Disposition Among Patients Admitted for Heart Failure in the United States. Am J Cardiol. 2017 Sep 1;120(5):817-824. doi: 10.1016/j.amjcard.2017.05.058. Epub 2017 Jun 15. PMID 28705376
- [Background] Khan H, Greene SJ, Fonarow GC, Kalogeropoulos AP, Ambrosy AP, Maggioni AP, Zannad F, Konstam MA, Swedberg K, Yancy CW, Gheorghiade M, Butler J; EVEREST Trial Investigators. Length of hospital stay and 30-day readmission following heart failure hospitalization: insights from the EVEREST trial. Eur J Heart Fail. 2015 Oct;17(10):1022-31. doi: 10.1002/ejhf.282. Epub 2015 May 9. PMID 25960401
- [Background] Sud M, Yu B, Wijeysundera HC, Austin PC, Ko DT, Braga J, Cram P, Spertus JA, Domanski M, Lee DS. Associations Between Short or Long Length of Stay and 30-Day Readmission and Mortality in Hospitalized Patients With Heart Failure. JACC Heart Fail. 2017 Aug;5(8):578-588. doi: 10.1016/j.jchf.2017.03.012. Epub 2017 May 10. PMID 28501521
- [Background] Reeves GR, Whellan DJ, Patel MJ, O'Connor CM, Duncan P, Eggebeen JD, Morgan TM, Hewston LA, Pastva AM, Kitzman DW. Comparison of Frequency of Frailty and Severely Impaired Physical Function in Patients >/=60 Years Hospitalized With Acute Decompensated Heart Failure Versus Chronic Stable Heart Failure With Reduced and Preserved Left Ventricular Ejection Fraction. Am J Cardiol. 2016 Jun 15;117(12):1953-8. doi: 10.1016/j.amjcard.2016.03.046. Epub 2016 Apr 6. PMID 27156830
- [Background] Sica DA, Muntendam P, Myers RL, Ter Maaten JM, Sale ME, de Boer RA, Pitt B. Subcutaneous Furosemide in Heart Failure: Pharmacokinetic Characteristics of a Newly Buffered Solution. JACC Basic Transl Sci. 2018 Feb 7;3(1):25-34. doi: 10.1016/j.jacbts.2017.10.001. eCollection 2018 Feb. PMID 30062191